CLINICAL TRIAL: NCT07009366
Title: Comparison of Methods of Weaning From Nasal CPAP in Preterm Infants: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DRRABIAZUK
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sudden weaning of NCPAP (Experimental): NCPAP was taken "off" entirely when the neonate met the "stability criteria" and remained on oxygen or room air via a headbox or incubator with an aim to stay off NCPAP.
  Interventions: Procedure: Sudden weaning of NCPAP
- Gradual Weaning with increasing the time off NCPAP (Experimental): The regimen adopted for this method was 1 hour off twice a day on the 1st day, then 2 hours off twice a day on the 2nd day, hence increasing the time off to 6 hours twice a day (or 12 hours per day), i.e., using a smaller period off. At this point, NCPAP was taken off completely.
  Interventions: Procedure: Gradual weaning with increasing the time off NCPAP
- Pressure weaning of NCPAP (Experimental): In this method the pressure was reduced in steps of 1 cm of H2O every 12 to 24 hours until 5 cm of H2O, and then if the child tolerated it well, NCPAP was removed, and the child was shifted to oxygen via incubator or room air according to the situation.
  Interventions: Procedure: Pressure weaning of NCPAP

INTERVENTIONS:
Procedure: Sudden weaning of NCPAP — NCPAP was taken "off" entirely when the neonate met the "stability criteria" and remained on oxygen or room air via a headbox or incubator with an aim to stay off NCPAP.
  Arms: Sudden weaning of NCPAP
Procedure: Gradual weaning with increasing the time off NCPAP — The regimen adopted for this method was 1 hour off twice a day on the 1st day, then 2 hours off twice a day on the 2nd day, hence increasing the time off to 6 hours twice a day (or 12 hours per day), i.e., using a smaller period off. At this point, NCPAP was taken off completely.
  Arms: Gradual Weaning with increasing the time off NCPAP
Procedure: Pressure weaning of NCPAP — In this method the pressure was reduced in steps of 1 cm of H2O every 12 to 24 hours until 5 cm of H2O, and then if the child tolerated it well, NCPAP was removed, and the child was shifted to oxygen via incubator or room air according to the situation.
  Arms: Pressure weaning of NCPAP

SUMMARY:
This study aimed to determine the efficacy of different NCPAP weaning strategies in pre-term infants presenting with respiratory distress, and ultimately establishing the best method to withdraw from NCPAP.

DETAILED DESCRIPTION:
Pakistan, as well as other developing countries, lacks data regarding the weaning protocol of NCPAP. Ascertaining the best weaning method that could facilitate a shorter duration on nasal CPAP and the least length of hospital stay is very much needed. Findings of this study would help clinicians to achieve better outcomes for the patients receiving nasal CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants
* Any gender
* Low birth weight
* Gestational ages between 28 to below 37 weeks
* Presented with respiratory distress
* Neonates with radiological findings suggestive of respiratory distress, congenital pneumonia/sepsis, or transient tachypnea of the newborn (TTN)

Exclusion Criteria:

* Complex congenital abnormalities like diaphragmatic hernia, CNS malformations, intrapartum-related hypoxia, or congenital heart disease.
* Intraventricular hemorrhage grade III or IV or low APGAR scores (<4 or 5 at 5 minutes)

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Successful weaning | 4 days
  Weaning was considered as successful in the absence of pronounced retractions, tachypnea, or episodes of apnea and if there was no requirement for ventilator support after cessation of NCPAP support.

SECONDARY OUTCOMES:
Comparison of total days on NCPAP | 4 days
  Total days on NCPAP for the three weaning strategies were measured from the start of NCPAP to the removal of NCPAP
Hospital stay | 25 days
  Total days of hospital stay were measured from the admission to discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Asif, Principal Investigator — Ziauddin University Karachi; Heena Rais, FCPS, Study Director — Ziauddin University Karachi
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.